CLINICAL TRIAL: NCT05785273
Title: Intraoperative Assessment of Analgesic Depth During General Anesthesia With Dexmedetomidine-remifentanil Infusion. A Pilot Study
Brief Title: Analgesic Depth Evaluation During General Anesthesia With Dexmedetomidine-remifentanil Infusion. A Pilot Study
Status: Completed | Type: Observational
Sponsor: Università degli Studi di Brescia (Other)
Collaborators: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Martino Stefanini, Principal investigator, Università degli Studi di Brescia
Other Study IDs: UBrescia NP 3675
Record Dates: First submitted 2023-02-20; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Analgesia; Anesthesia
Keywords: Dexmedetomidine; Pupil; Nociception; Opioid sparing
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dexmedetomidine: Patient undergoing general anesthesia receving initial administration of dexmedetomidine loading dose of 0.5-1 μg/kg (ADJUSTED weight) over 15 minutes. After intubation maintenance of general anesthesia is administrated with desflurane or sevoflurane (MAC 0.6 - 1, according to Bispectral Index (BIS) or Patient State Index (Psi)), dexmedetomidine (0.2- 0.4 μg/kg/h (Lean Body Weight)) with constant infusion rate unless hypotension or bradycardia not responsive to standard treatments (filling, atropine, ephedrine, ethylephrine) occurred, and remifentanil (0.02 - 0.2 μg/kg/min (LBW)) based on clinical and instrumental assessment (Heart Rate, Blood Pressure, BIS or Psi).
  Interventions: Device: Pupillometer
- No Dexmedetomidine: Patients in this group receive an eventual premedication with benzodiazepines according to anaesthesiologist assessment and patient condition. After intubation general anesthesia is administrated with inhaled (desflurane or sevoflurane; MAC 0.6 - 1) or intravenous (propofol) anesthetics (according to BIS or Psi) and remifentanil (0.02 - 0.2 μg/kg/min (LBW) based on clinical and instrumental assessment (HR, BP, BIS or Psi)).
  Interventions: Device: Pupillometer

INTERVENTIONS:
Device: Pupillometer — 1st pupil evaluation between induction of general anesthesia and onset of surgery. After incision, at least 3 pupil evaluations are performed. Measurements are spaced 15 minutes apart and also taken at least 10 minutes after any variation in drugs dosage

SUMMARY:
The aim of this study is to verify the feasibility of an evaluation of the depth of analgesia during an opioid sparing anesthesia (OSA) carried out with continuous infusion of dexmedetomidine in addition to general multimodal anesthesia trough an instrumental pupillary evaluation.

DETAILED DESCRIPTION:
In recent years, different strategies have been proposed to reduce opioid use during the perioperative period, i.e., the so-called OFA (opioid free anesthesia) or OSA (opioid sparing anesthesia), in order to reduce some opioid-related side effects with equivalent intraoperative analgesia compared to opioid-based anesthesia.

Dexmedetomidine is a highly selective α2-agonist, with sedative and pain-relieving effects. The use of perioperative dexmedetomidine seems to reduce intraoperative opioid and hypnotic consumption, postoperative pain intensity and postoperative opioid use.

A dexmedetomidine-based protocol for anesthesia in obese patients was introduced in our department towards the end of 2018. All patients undergoing bariatric surgery have been treated with a premedication of dexmedetomidine and a steady infusion of dexmedetomidine as an opioid-savings adjuvant during general anesthesia. In this context, the amount of fentanyl (induction of anesthesia) and remifentanil (maintenance of anesthesia) has been reduced empirically and clinically.

Traditionally, during general anesthesia, the level of nociception is indirectly assessed by observing heart rate, blood pressure and surgical steps. In recent years, new indicators have been proposed to obtain an objective and standardized nociception assessment. Pupillary dilation reflex (PDR) can be related to both painful stimulation and analgesic depth, but not to neuromuscular blockade or hypnotic drug administration. Recently, another rating scale for nociception has been proposed: the PPI (pupillary pain index). This index is based on tetanic stimulation of increasing intensity delivered by two skin electrodes placed on the forearm, evaluating the PDR at each stimulus. A PPI from 1 to 3, from 4 to 6, or from 7 to 9 describes a numbed PDR and deep analgesia, a medium PDR and suboptimal analgesia and a highly reactive PDR and uncontrolled pain, respectively.

The investigators proposal is to study the feasibility of an evaluation of the nociception during an Opioid Sparing Anesthesia (OSA), with continuous infusion of dexmedetomidine and remifentanil, vs "traditional" anesthesia without adjuvant, using the PPI as an indicator of nociception.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent open surgery involving at least one surgical incision of more than 5 cm
* use of remifentanil as an intravenous analgesic.

Exclusion Criteria:

* implanted pacemaker or ICD
* ophthalmological comorbidities
* chronic opioid use
* peripheral neuropathy
* continuous infusion of adjuvant drugs other than dexmedetomidine
* epidural analgesia or loco-regional block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent no-laparoscopic surgery involving at least one surgical incision of more than 5 cm with remifentanil as an intravenous analgesic.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of study protocol | 6 months
  Number of patients enrolled and number of pupillary evaluation during anesthesia

SECONDARY OUTCOMES:
Depth of analgesia | Intraoperative
  depth of intraoperative analgesia with PPI (pupillary pain index). A PPI from 1 to 3, from 4 to 6, or from 7 to 9 describes a numbed PDR and deep analgesia, a medium PDR and suboptimal analgesia and a highly reactive PDR and uncontrolled pain, respectively.
Intra-operative opioid consumption | Intraoperative
  total consumption of remifentanil (μg/kg/min - Lean Body Weight)
Incidence of side effects | Intraoperative
  incidence of perioperative side effects, PONV and post-operative intolerable pain in the first 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Frank A Rasulo, MD, Study Director — Università degli Studi di Brescia
Locations (1):
- ASST Spedali Civili, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grape S, Kirkham KR, Frauenknecht J, Albrecht E. Intra-operative analgesia with remifentanil vs. dexmedetomidine: a systematic review and meta-analysis with trial sequential analysis. Anaesthesia. 2019 Jun;74(6):793-800. doi: 10.1111/anae.14657. Epub 2019 Apr 5. PMID 30950522
- [Background] Sabourdin N, Barrois J, Louvet N, Rigouzzo A, Guye ML, Dadure C, Constant I. Pupillometry-guided Intraoperative Remifentanil Administration versus Standard Practice Influences Opioid Use: A Randomized Study. Anesthesiology. 2017 Aug;127(2):284-292. doi: 10.1097/ALN.0000000000001705. PMID 28719527
- [Background] Kim JH, Jwa EK, Choung Y, Yeon HJ, Kim SY, Kim E. Comparison of Pupillometry With Surgical Pleth Index Monitoring on Perioperative Opioid Consumption and Nociception During Propofol-Remifentanil Anesthesia: A Prospective Randomized Controlled Trial. Anesth Analg. 2020 Nov;131(5):1589-1598. doi: 10.1213/ANE.0000000000004958. PMID 33079883
- [Derived] Stefanini M, Cagnazzi E, Calza S, Latronico N, Rasulo FA. Feasibility of the pupillary pain index as a guide for depth of analgesia during opioid-sparing anesthesia with continuous infusion of dexmedetomidine. J Anesth Analg Crit Care. 2023 Aug 14;3(1):27. doi: 10.1186/s44158-023-00112-8. PMID 37580838